CLINICAL TRIAL: NCT05313945
Title: Multicenter, Randomized, Controlled Trial Evaluating Patient Satisfaction After Passive Bladder Catheter Removal Following Urological Surgery Compared to Active Removal by a Nurse
Brief Title: Evaluation Patient Satisfaction After Passive Bladder Catheter Removal Compared to Active Removal
Acronym: IDESONDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_0171
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Urologic Diseases
Keywords: bladder catheter
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive indwelling urinary catheter removal (Experimental): The passive indwelling urinary catheter removal takes place due to gravity.
  Interventions: Procedure: Passive indwelling urinary catheter removal
- Manual indwelling urinary catheter removal (Active Comparator): The manual indwelling urinary catheter removal takes place by manual traction by a nurse.
  Interventions: Procedure: Active indwelling catheter removal by a nurse

INTERVENTIONS:
Procedure: Passive indwelling urinary catheter removal — After washing the patient's perineal area with water and mild soap, the nurse deflates the indwelling urinary catheter balloon and instructs the patient to take a shower (standing).
  During this time, the catheter will fall under gravity.
  Arms: Passive indwelling urinary catheter removal
Procedure: Active indwelling catheter removal by a nurse — After washing the patient's perineal area with water and mild soap, the nurse deflates the balloon and removes the catheter from the urethra by manual traction.
  Arms: Manual indwelling urinary catheter removal

SUMMARY:
In usual practice, the removal of the bladder catheter is performed by a nurse a few days after the surgery. The nurse deflates the balloon and removes the catheter from the urethra by manual traction. To date, there are no solid data on the impact of passive catheter removal on patient satisfaction.

It is therefore necessary to estimate the effect on patient satisfaction of active catheter removal by a nurse versus passive catheter removal under gravity. The effect on pain and anxiety will also be compared between the two techniques. The methodology used was that of an open-label randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years old
2. With an indwelling urinary catheter placed after any of the following procedures:

   A uro-endoscopic surgery from the list below:
   * Endoscopic prostate resection (or transurethral prostate resection).
   * Laser prostate enucleation
   * Prostate thermotherapy by radiofrequency
   * A high-intensity focused ultrasound treatment for prostate cancer
   * Cervico-prostatic incision or internal urethrotomy
   * Endoscopic/Transurethral Resection of Bladder Tumor (TURBT)
   * Surgical treatment of bladder stones, ureter stones (rigid ureteroscopy) and kidney stones (flexible ureteroscopy with laser stone fragmentation)
3. Patient who has given written consent to participate

Exclusion Criteria:

1. Patient who is unable to perform intimate hygiene alone in a standing position
2. Patient with a painful genital lesion
3. Patient with an extended pelvic pathology
4. Need to remove the indwelling urinary catheter at the patient's home instead of hospital
5. Patient under guardianship or curator
6. Patient unable to understand the objectives of the study or unwilling to comply with postoperative instructions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction score | Within one hour after indwelling urinary catheter removal at day 0
  Patient satisfaction score using a numerical rating scale (NRS) from the minimum value 0 (The worse score) to the maximum value 10 (The better Score)

SECONDARY OUTCOMES:
The pain experienced by patients | Prior to catheter removal (within 30 minutes before the start of the procedure) and in the immediate aftermath (within one hour after the removal of the catheter)
  The pain experienced by patients will be measured using a numerical scale (EN) ranging from the minimum value 0 (The better score) to the maximum value 10 (The worse Score)
The anxiety experienced by patients | Prior to catheter removal (within 30 minutes before the start of the procedure) and in the immediate aftermath (within one hour after the removal of the catheter)
  The anxiety experienced by patients will be measured using a numerical scale (EN) ranging from the minimum value 0 (The better score) to the maximum value 10 (The worse Score)
Patient satisfaction | at Day 0, at Day 2, at Day 15
  Patient satisfaction will be evaluated using a satisfaction questionnaire without score
Patient satisfaction | at Day 2, at Day 15
  Patient satisfaction score using a numerical rating scale (NRS) from the minimum value 0 (The worse score) to the maximum value 10 (The better Score)

CONTACTS AND LOCATIONS:
Overall Officials: Camille BENETON, Nurse, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - CHU Grenoble, Grenoble
  - Hôpita Edouard Herriot, Lyon